CLINICAL TRIAL: NCT03764267
Title: Monitored Anesthesia Care Using Remifentanil and Ketofol Results in a Superior Quality of Recovery Compared With Total Intravenous Anesthesia in Ambulatory Breast Augmentation
Brief Title: MAC vs TIVA Ambulatory Breast Augmentation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Wahba bakhet, Lectrure of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ainshamsuni-MAC-wbakhet
Record Dates: First submitted 2018-12-01; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases | interventions — Remifentanil; Lidocaine; Anesthetics, General

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- remifentanil (Active Comparator): MAC group
  Interventions: Drug: Remifentanil
- general anesthetic (Active Comparator): TIVA group
  Interventions: Drug: general anesthetic

INTERVENTIONS:
Drug: Remifentanil — Five minutes before infiltration of the local anesthestic by the surgeon, patients received an initial maintenance infusion of remifentanil 0.1 µg/kg/min and ketofol mixture 0.3 ml/kg (propofol 25 µg /kg/min and ketamine 10 µg/kg/min). ketofol mixture was prepared in a ratio of 1:2.5 (100 mg ketamine 2 mL (100 mg), propofol 1% 25 mL (250 mg), and glucose 5% 23 ml, total volume of 50 ml, each ml contain 2 mg ketamine + 5 mg propofol).
  Throughout the surgery, titration of the infusion rate of the remifentanil and ketofol were indicated by vital signs and expression of pain
  Other Names: lidocaine, ropivaicaine
  Arms: remifentanil
Drug: general anesthetic — general anesthetic was induced with a bolus dose of remifentanil (1 ug/kg over 30 second) and propofol (2 mg/kg) followed by insertion of a laryngeal mask airway (LMA). After the induction of anaesthesia and securing the airway, patient' lungs were ventilated with volume controlled ventilation, 50% oxygen/air mixtures in a circle system. .Anesthesia was maintained with remifentanil (0.5 ug/ kg/ min) and propofol (5 mg/kg/h). Remifentanil and propofol titrated to keep heart rate and the blood pressure within 20% of the baseline values and maintain BIS between 40 and 60, respectively. Patient movements were treated with additional i.v. bolus doses of remifentanil 0.5 ug/kg
  Other Names: total intravenous anesthesia
  Arms: general anesthetic

SUMMARY:
hypothesis: the combination of LA with remifentanil and ketofol [monitored anesthesia care (MAC)] for ambulatory breast augmentation may result in results in better QoR on day of surgery as compared with total i.v. anesthesia (TIVA) . The purpose of this study was to compare the QoR after MAC using remifentanil and ketofol with TIVA during ambulatory breast augmentation .

DETAILED DESCRIPTION:
Breast augmentation surgery is commonly performed on an ambulatory basis under under general anesthesia (GA) with propofol and remifentanil or local anesthesia (LA). Although surgeons perform this operation comfortably under GA, Patients have anxiety and fear of complications due to GA. In addition, they expect a good postoperative quality of recovery (QOR) including ability to resume common activities (work and daily activities) without suffering from moderate to severe pain.

The LA is advantageous over GA in that airway instrumentation is not necessary, favorable recovery profile, decrease postoperative pain and vomiting, increase patient satisfaction and decrease the cost . However, patient anxiety or pain often leading to conversion of LA to GA, which suggests the concomitant use of i.v. sedatives and analgesics as a supplement to LA.

The combination of remifentanil and ketofol (propofol, ketamine) for sedation during regional anesthesia and LA has been shown to be a safe, effective technique, capable of maintains adequate analgesia with conscious sedation, haemodynamic stability, and achieves lower incidence of postoperative nausea and vomiting with shorter recovery times.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II

Exclusion Criteria:

* ASA III

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | 24 hours postoperative
  Quality of recovery-40 (QoR-40) questionnaire, which includes five general quality of life dimensions: physical independence (5 items), pain (7 items), .emotional state (9 items), psychological support (7 items), and physical independence (5 items). Each item was graded with a 5-point score: none of the time, some of the time,usually, most of the time and all of the time. The total score on the QoR- 40 questionnaire ranges from 40 to 200 representing, respectively, extremely poor to excellent

SECONDARY OUTCOMES:
Recovery room readiness times | 24 hours postoperative
  minutes
home readiness times | 24 hours postoperative
  minutes
adverse events | 24 hours postoperative
  vomiting

IPD SHARING:
Plan to Share IPD: Undecided